CLINICAL TRIAL: NCT03278886
Title: Pilot Study of Opioid-receptor Antagonists to Reduce Pain and Inflammation Among HIV-Infected Persons With Alcohol Problems
Brief Title: St. PETERsburg Pain and Alcohol Intervention With Naltrexone and Nalmefene
Acronym: PETER PAIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-36491; UH2AA026193 (NIH)
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: HIV Infection; Alcohol Use; Pain
Keywords: Alcohol Use; Pain; HIV; Low-dose naltrexone; Nalmefene
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Pain | interventions — Naltrexone; nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose naltrexone (Experimental): Participants randomized to this group will receive low dose naltrexone (4.5 mg) for 8 weeks.
  Interventions: Drug: Low dose naltrexone
- Nalmefene (Experimental): Participants randomized to this group will receive nalmefene (18 mg) for 8 weeks.
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Low dose naltrexone — 4.5 mg of low dose naltrexone taken once daily for 8 weeks
  Arms: Low dose naltrexone
Drug: Nalmefene — 18 mg of nalmefene taken once daily for 8 weeks
  Arms: Nalmefene

SUMMARY:
This study is a randomized controlled trial (RCT) to assess the feasibility, tolerability, and safety of using opioid receptor antagonists (naltrexone and nalmefene) to treat pain among HIV-infected persons with heavy alcohol use and chronic pain.

DETAILED DESCRIPTION:
Pain is a common co-morbidity for HIV-infected patients. Prevalence studies suggest that, on average, half of all HIV-infected persons suffer pain. Chronic pain can lead to heavy alcohol use among HIV-infected persons, which may in turn be a barrier to treatment/control of HIV and contribute to spread of HIV. Thus there is an urgent need to address pain among persons with HIV. Opioid receptor antagonists such as naltrexone and nalmefene, which are licensed for treatment of alcohol use disorders, show promise as being effective and safe treatments for chronic pain among persons with HIV. This study will pilot test novel pharmacotherapies (opioid receptor antagonists) to improve chronic pain among HIV-infected heavy drinkers. The specific aims of the research is to assess the feasibility, tolerability and safety of using opioid receptor antagonists (low-dose naltrexone and nalmefene) to treat pain among HIV-infected persons with heavy alcohol use and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HIV-positive
* Chronic pain (present ≥3 mo) of moderate to severe intensity
* Heavy drinking past year (Based on NIAAA criteria: > 14 standard drinks per week/ > 4 drinks in a day for men; > 7 drinks in the past week/ > 3 drinks in a day for women)
* If female, negative pregnancy test and willing to use adequate birth control
* Provision of contact information for 2 contacts to assist with follow-up
* Stable address within 100 kilometers of St. Petersburg
* Possession of a telephone (home or cell)
* Able and willing to comply with all study protocols and procedures

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment resulting in inability to provide informed consent based on research assessor (RA) assessment
* Known active TB or current febrile illness
* Breastfeeding
* Uncontrolled psychiatric illness (such as active psychosis) (i.e., answered yes to any of the following: past three month active hallucinations; mental health symptoms prompting a visit to the ED or hospital)
* History of hypersensitivity to naltrexone, nalmefene, or naloxone
* Current use (past week) of illicit or prescribed opiates as documented by either self-report or positive urine drug test
* Unwilling to abstain from opiates during the treatment period
* Current use of neuroleptics
* History of seizure disorder
* Known liver failure
* ALT/AST levels >5x normal
* History of Raynaud's Disease
* Planned surgeries in the next three months
* Enrolled in another HIV and/or substance use medication intervention study
* Taking naltrexone in the past 30 days
* Taking nalmefene in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Samet, MD, MA, MPH, Principal Investigator — Boston University/Boston Medical Center
Locations (1):
- First St. Petersburg Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
All data from the study will be placed into the URBAN ARCH repository.
URL: http://www.urbanarch.org

REFERENCES:
- [Derived] Bendiks S, Cheng DM, Blokhina E, Vetrova M, Verbitskaya E, Gnatienko N, Bryant K, Krupitsky E, Samet JH, Tsui JI. Pilot study of tolerability and safety of opioid receptor antagonists as novel therapies for chronic pain among persons living with HIV with past year heavy drinking: a randomized controlled trial. AIDS Care. 2023 Aug;35(8):1191-1200. doi: 10.1080/09540121.2021.1896663. Epub 2021 Mar 7. PMID 33682527
- See also: URBAN ARCH, a member of NIAAA CHAART (Consortiums for HIV/AIDS & Alcohol Research Translation) initiative, conducts and disseminates interdisciplinary research on how alcohol impacts people with HIV and develops interventions to reduce related outcomes. — http://www.urbanarch.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Naltrexone | Nalmefene
Started | 8 | 3
Completed | 8 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Naltrexone | Nalmefene | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (7.46) | 35.7 (1.09) | 37.8 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 8 | 3 | 11
Education (9 grades or more) [Count of Participants; unit: Participants] | 8 | 3 | 11
Married/Living with partner/In long-term relationship [Count of Participants; unit: Participants] | 5 | 3 | 8
At risk drinking based on NIAAA criteria [Count of Participants; unit: Participants] — At risk drinking defined as >14 standard drinks per week/ > 4 drinks in a day for men; > 7 drinks in the past week/ > 3 drinks in a day for women.
  Participants | 2 | 1 | 3
Lifetime opioid use [Count of Participants; unit: Participants] | 5 | 3 | 8
Past 30 day opioid use [Count of Participants; unit: Participants] | 0 | 0 | 0
Pain severity [Median (Inter-Quartile Range); unit: units on a scale] — Scale of 1-10 with higher numbers indicating greater levels of pain
  units on a scale | 3.0 [2.1 to 4.5] | 4.5 [4.0 to 5.5] | 3.3 [2.5 to 5.5]
Pain interference [Median (Inter-Quartile Range); unit: units on a scale] — Scale of 1-10 with higher numbers indicating greater levels of pain
  units on a scale | 2.5 [2.0 to 6.7] | 5.6 [4.1 to 7.9] | 4.1 [2.1 to 6.1]
Cold pain threshold [Median (Inter-Quartile Range); unit: seconds] — Measured as number of seconds to the initial perception of pain during cold-pressor test
  seconds | 9.5 [7.9 to 13.5] | 10 [3.6 to 13.5] | 10 [6.7 to 13.1]
Cold pain tolerance [Median (Inter-Quartile Range); unit: seconds] — Measured as seconds until withdrawal of hand during cold-pressor test
  seconds | 19.3 [16.5 to 22.8] | 22 [8.2 to 22.5] | 19.5 [14 to 22.5]

OUTCOME MEASURES:

1. Primary Outcome: Medication Tolerability Measured Via a 0-100 Visual Analog Scale
Description: Medication tolerability will be measured via a 0-100 visual analog scale. Participants will be asked to indicate on a scale of 0-100, how well they have tolerated the study medication with 0 anchored as "cannot tolerate at all" and 100 as "tolerate perfectly well." Higher numbers will be indicative of higher tolerability of the medication.
Time Frame: Primary endpoint at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
score on a scale | 90.7 (22.4) | NA (NA) — All participants randomized to this arm discontinued study medication due to side effects. At 8-weeks, no participants in this arm were taking the study medication, so a tolerability score was not assessed.

2. Secondary Outcome: Change in Alcohol Use Defined as a Change in the Mean Number of Grams of Pure Ethanol Consumed Per Day From Baseline to 8 Weeks
Description: Measured via 30 Day Alcohol Use Timeline Follow Back Method
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: grams of ethanol
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
grams of ethanol | 5.5 (10.1) | -6.83 (9.7)

3. Secondary Outcome: Treatment Discontinuation Defined as Patient Self-report of Stopping Medication Anytime During the Treatment Period
Description: Measured via one question asking participants if they had discontinued medication since their last visit. Assessed at 4 and 8 week study visits.
Time Frame: 4 weeks, 8 weeks
Measure: Number; unit: treatment discontinuations
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
treatment discontinuations
  4-Weeks | 1 | 1
  8-Weeks | 1 | 2

4. Secondary Outcome: Adherence to Medication Defined as Self-report of Percentage of Study Medication Taken in the Past Two Weeks
Description: Measured by participants' drawing a line on a a Visual Analog Scale, which ranges from 0 to 100. Higher numbers indicate higher adherence to study medication.
Time Frame: Endpoint at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
score on a scale | 87.5 (35.4) | 0 (0)

5. Secondary Outcome: Number of Participants With Adherence Assessed Via Riboflavin in the Urine Confirming Adherence
Description: Measured through visual inspection of the urine for the presence or absence of riboflavin using ultraviolet (UV) light at the long wave setting (33 mm) in a room with low ambient light.
Time Frame: Endpoint at 8 weeks
Measure: Number; unit: participants
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
participants | 1 | 0

6. Secondary Outcome: Reported Side Effects Using a Symptom Checklist, Plus an Open-ended Question
Description: Measured via a 16-item symptom checklist with the option for participants to report any experienced side effects not on the checklist. Side effect severity is rated by trained research assessors. The checklist is asked at 2, 4, 6, and 8-week study visits.
Time Frame: 2 weeks, 4 weeks, 6 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: number of side effects
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
number of side effects
  2-Weeks | 1.5 (1.6) | 4.5 (6.4)
  4-Weeks | 1.3 (1.2) | 1.5 (2.1)
  6-Weeks | 0.9 (1.0) | 1.5 (2.1)
  8-Weeks | 0 (0) | 0 (0)

7. Secondary Outcome: Medication Satisfaction Defined as a Score From 0-100 Measured Via the Treatment Satisfaction Questionnaire for Medication (TSQM), With Higher Scores Corresponding to Higher Treatment Satisfaction.
Description: Measured via using the 14-item Treatment Satisfaction Questionnaire, which consists of 14 items that result in four domains: Effectiveness, Side Effects, Convenience and Global Satisfaction. Higher scores indicate greater satisfaction with medication. Assessed at 4 and 8 week study visits.
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
score on a scale
  4-Weeks | 47.3 (24.4) | 3.6 (5.1)
  8-Weeks | 47.3 (21.9) | 3.6 (5.1)

8. Secondary Outcome: Severe Hepatotoxicity Defined as AST/ALT >10X the Level of Normal
Description: Aminotransferase levels (AST/ALT) are tested to look for severe hepatotoxicity defined as AST/ALT > 10 times the level of normal.
Time Frame: Endpoint at 8 weeks
Measure: Number; unit: participants
Arm/Group | Low Dose Naltrexone | Nalmefene
Number analyzed (Participants) | 8 | 2
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the 8-week treatment period.
Arm/Group | Low Dose Naltrexone | Nalmefene
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/3
Other Adverse Events (participants affected / at risk) | 3/8 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Naltrexone (N=8) | Nalmefene (N=3)
Body injury during fight (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Naltrexone (N=8) | Nalmefene (N=3)
Agitation (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams/nightmares (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep problems (Psychiatric disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03278886/Prot_SAP_000.pdf